CLINICAL TRIAL: NCT00283348
Title: New Strategies for Non-invasive Detection of Chronic Allograft Nephropathy
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: Cell 500
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Chronic Rejection
Keywords: Renal Transplantation; Immunosuppression; Chronic Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to help researchers find out more about a condition called "Chronic Allograft Nephropathy" (CAN). CAN is a complication that sometimes occurs after kidney transplantation and affects the function of the transplanted kidney. It is hoped that by studying blood, urine, and tissue samples of kidney transplant patients, new ways of diagnosing and treating CAN may be found.

DETAILED DESCRIPTION:
We hypothesize that patients with CAN will manifest different patterns of gene expression profiling (compared with non-CAN controls), detectable in peripheral blood mononuclear cells (PBMCs) and urine cells. By studying differences that exist in peripheral blood or in the graft and its local environment (urine samples), informative biomarkers may be discovered to improve treatment programs.

Specific Aims:

AIM 1: To investigate the genes involved in the molecular mechanism that characterize CAN in kidney transplant recipients, we will study gene expression in kidney biopsy samples from patients with CAN. For comparison analysis, we will study gene expression profiling in normal kidney biopsies (Control Group 1).

AIM 2: To determine whether there is a role for assessing peripheral blood mononuclear cell (PBMC) and urine cell gene expression patterns as a means of measuring the immunologic and clinical status of kidney transplant recipients, we will compare gene expression profiles among PBMC, urine and biopsy samples.

AIM 3: To establish the clinical utility of the set of markers resulting from AIMS 1 and 2 in the diagnostic of CAN, we will use "real time"(RT)-PCR in PBMC and urine samples employing a limited panel of markers in an independent group of patients.

AIM 4: To study the role of the pre-established panel of molecular markers in the early detection of CAN in patients receiving mycophenolate mofetil (MMF) as immunosuppressive treatment, we will study urine and PBMC samples from patients more than 12 months post-transplantation, with normal creatinine, and proteinuria.

Background and Significance:

Chronic allograft nephropathy (CAN) is a devastating complication of kidney transplantation that is responsible for a significant proportion of graft loss (1-5). Although currently available immunosuppressive therapy is increasingly effective against acute rejection of a transplanted organ, chronic rejection (CR) remains difficult to treat. Nevertheless, a relevant proportion of patients with CR of a kidney transplant maintain satisfactory organ function for a long time. CAN is characterized by a progressive decline in kidney function, which is not attributable to a specific cause (6-8). CAN is a poorly known complex process resulting from as yet undefined etiology with both immune and non-immune components (8). Alloantigen-dependent causes of CAN include acute rejection episodes, particularly multiple, late, or vascular acute rejection episodes (9-13). With the use of a new immunosuppressive regimen, the frequency of acute rejection episodes has become reduced, which may possibly have an influence on future development of CAN. However, donor antigen-independent factors also play a role in the occurrence and progression of CAN. This includes donor-related factors such as donor age and number of mismatch, which have an impact on late graft outcome (13). Donation-related circumstances, such as prolonged cold ischemia time, are associated with delayed graft function and related to poor late renal transplant results.

Recipient related factors may also act as co-factors contributing to an accelerated deterioration of the functional units in the kidney, including vascular, of renal arteries and a subsequent relative hypoxia of the kidney, frequently leading to interstitial fibrosis. Interestingly, many of the pathways involved in chronic injury and fibrosis are regulated very early in the course of the injury, when the downstream effects of these alterations are still not evident by pathology.

The histopathologic features of CAN can be characterized by proliferative changes of the vascular wall, in which smooth muscle cells and parenchymal cells proliferate, leading to a narrowing of renal arteries, which may contribute to a relative hypoxia of the tissue. Subsequently, fibroblasts will contribute to fibrotic scarring in the vascular wall. CAN is also characterized by the occurrence of fibrosis in the interstitial tissue along with tubular atrophy (14). The glomeruli are also often affected by various degrees of glomerulosclerosis. An inflammatory infiltrate is frequently found and consists of invading lymphocytes and monocytes-macrophages into virtually all affected compartments of the kidney. The inflammatory infiltrate observed in CAN can be induced by both antigen-dependent and antigen-independent factors. These histopathologic changes can be graded according to the Banff system (14), which gives a score of the degree of CAN. These histopathologic changes act in concert, contributing to a gradual progression of renal allograft dysfunction.

Fundamental studies in solid organ transplantation have characterized specific functional roles for individual genes in the immunological cascade leading to organ rejection. Nevertheless, significant redundancy in the immune system is suggested by clinical variability in acute rejection outcomes, in the progression of chronic rejection, and by the potential to acquire graft tolerance. Underlying all of these complex systems are concordant expression and co-regulation of multiple genes in known and novel molecular pathways. Ascertaining their individual functions in adapting the effector response is now possible with gene expression profiling using microarrays. Although cDNA microarrays (large numbers of genes represented by complementary DNAs or oligonucleotides immobilized onto microscope slides or silicon chips) were successfully used to profile gene expression in cancer (15,16,17,18,19), their impact in transplantation research has so far been relatively modest.

I suggest that the highlighted section be deleted, or at least placed in parentheses. It makes the sentence very difficult to understand, though I know it is meant to clarify.

There is accumulating evidence that non-invasive immune monitoring may be useful in the early period after renal transplant (20,21), particularly with regard to predicting the presence of acute rejection. It is less clear whether chronic allograft nephropathy (CAN) is also associated with consistent changes in peripheral blood or urine cells.

Moreover, current methods of diagnosing allograft dysfunction are inadequate for detecting the significant organ damage that occurs prior to the establishment of clinical manifestations. The development of assays or novel technologies that will allow detection of allograft dysfunction/rejection, monitor responses to therapy, and predict long-term outcomes is vital for the success of transplantation.

In this project we propose to establish the molecular markers that characterize CAN using gene expression profiling in kidney biopsies of patients with CAN and to relate these findings with the profiles in PBMC and urine samples from the same patients. In addition, we will establish and validate (in a independent group of patients) the clinical utility of a limited set of molecular markers, resulting of the microarray analysis, using RT-PCR.

V. Statistical Analysis:

Data Security Plan Kidney tissue, PBMC and urine from kidney transplant patients with or without CAN will be studied. A Secure Data Base containing all the demographic information for the patients will be kept at the Virginia Commonwealth University, but patient identifiers will be removed and a study number assigned to each patient. The tissues required will include kidney biopsies only from patients with CAN.

Human Subjects:

A. Description and Research Materials Kidney tissues will be obtained with informed consent from patients with clinical suspicion of CAN (at least 15 patients). Tissue samples (needle biopsies) will be snap-frozen in liquid nitrogen within 5 minutes after excision and shipped under appropriate conditions, on dry ice, to maintain specimen integrity. All samples will be submitted for pathological evaluation, and a pathology report and clinical summary will be sent with the samples in all cases in a manner insuring patient confidentiality by removing patient identifiers and labeling with the assigned patient number.

Peripheral blood and urine samples (1-2 tbs) will be obtained from patients at the biopsy time. Kidney biopsies will be obtained with informed consent from normal kidneys at transplantation (needle biopsy from donor kidney, N=10).

Peripheral blood and urine samples will be collected monthly during 1 year with informed consent from kidney transplant patients with diagnostic of CAN confirmed by biopsy. As Control Group, stable long-term transplant patients (more than 12 months post-TX) with creatinine levels <1.6 mg/dL, and proteinuria less than 500mg/24hs, will be studied. (You may want to give an estimated number of patients to be included in the Control Group) All practices dealing with human subjects will be performed according to the ethical guidelines of the Institutional Review Board for the Protection of Human Subjects of the Virginia Commonwealth University.

Recruitment Plan Patients seen at VCU Hume-Lee Transplant Clinic who qualify according to the inclusion/exclusion criteria will be asked to participate in this study.

B. Potential Risks When blood is drawn there is a risk of bruising, bleeding, swelling or infection at the site where the blood is drawn.

Kidney biopsies can be painful where the needle enters the body, and a bruise can form. Bleeding can occur where the needle is inserted in to the kidney. Blood can appear in the urine.

Every effort will be made to maintain confidentiality. All identifying information will be kept in a secure data bank with access limited to research personnel.

C. Risk Reduction The tissue being obtained upon tissue biopsy is part of the sample that would be obtained for diagnostic purposes and not specifically for this protocol. The blood samples will be obtained at the same time as venous access is already in place. A urine sample will be collected prior to the biopsy.

All staff members handling tissue, PBMC and urine samples have been trained and are qualified to safely handle HCV infected tissue.

D. Risk/Benefit Because this is not a treatment study, there are no specific risks to the study subjects. CAN will be diagnosed and treated in the same way, whether or not they participate in the study. There is no guarantee that patients will benefit from participation in this study. The knowledge gained may be invaluable in the future particularly for diagnosing of CAN.

D. Compensation Plan Subjects will not be compensated for their participation in this study. E. Consent Issues Patients who meet study requirements will be consented.

ELIGIBILITY:
Inclusion Criteria:

* Received primary kidney transplant Diagnosis of Chronic Allograft Nephropathy Stable immunosuppression for one month prior to entry

Exclusion Criteria:

* Serious comorbidity Pregnancy Retransplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Diagnosis of Chronic Allograft Nephropathy at VCUHS Clinic
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Maluf, MD, Principal Investigator — Virginia Commonwealth University; Valeria Mas, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- VCU Health System, Richmond, Virginia, United States